CLINICAL TRIAL: NCT06079892
Title: Evaluation of Radiofrequency Efficiency in the Treatment of Hemorrhoid Pathology
Brief Title: Hemorrhoid Radiofrequency
Acronym: RFH
Status: Recruiting | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: 647-AAM-RFH
Record Dates: First submitted 2023-10-03; First posted 2023-10-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Hemorrhoid Prolapse
Keywords: radiofrequency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: radiofrequency — haemorrhoidal removal using radiofrequency

SUMMARY:
Triapedicular haemorroidectomy is currently the gold standard in haemorrhoidal pathology. Minimally invasive surgical techniques now play an important role in the haemorrhoidal management algorithm, particularly for less advanced stages of the disease. Among these techniques, radiofrequency is one of the most recent and is gradually gaining ground. It involves applying a radiofrequency current to the internal haemorrhoidal tissue in order to induce its involution.

The literature has shown that this technique leads to symptomatic improvement in over 60% of cases and a high satisfaction rate, even though some patients still seem to have haemorrhoidal symptoms postoperatively.

The aim of this study is to evaluate the efficacy of this technique in patients with haemorrhoidal pathology operated on at our centre, using "hard" criteria which are thought to be more rigorous ("cure" rather than "improvement").

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Presence of haemorrhoidal pathology
* Patient operated on between March 2017 and March 2023, using the radiofrequency technique
* French-speaking patient

Exclusion Criteria:

* ano-perineal involvement in Crohn's disease
* perianal fistula
* non-quiescent IBD
* radiation-induced rectitis
* psychiatric pathology.
* under guardianship or curatorship
* deprived of liberty
* under court protection
* Patient objecting to the use of his/her data for this research

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient suffering for Haemorroidal pathology and requiring a removal procedure to whom a Radiofrequency procedure was performed
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of radiofrequency treatment efficiency | 3 months post procedure
  Assessement of the procedure efficiency on prolapsus (using Goligher Score) and bleeding (using Haemorrhoidal bleeding score).
  Procedure is considered efficient when Goligher Score =1 AND HBS = 0

SECONDARY OUTCOMES:
Measurement of patient satisfaction after surgery | 3 months post procedure
  Patient will be asked :
  1. would you recommand this procedure to a friend ? (yes or no)
  2. Knowing your personnal outcome would you undergo the same procedure again ? (yes or no)
  Patients are considered satisfied by the procedure when they answered yes to at least one of the questions.
Incidence rate of procedure complication | 3 months post procedure
  incidence rate of haemorrhagic complication or acute urinary retention or other complication (such as post surgery abcess, localized infection, haematoma)
description of procedure complication | 3 months post procedure
Identification of predictive factor for success | 3 months post procedure
  pre-procedure parameters will be correlated with procedure success (Goligher Score =1 AND HBS = 0 after procedure) in order to identify which factors give a higher chance of success

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Hôpital Saint Joseph, Paris, France

IPD SHARING:
Plan to Share IPD: No